CLINICAL TRIAL: NCT04976257
Title: Pharmacokinetic Comparison of Selective Prostatic Arterial and Intravenous PSMA Radioligand Infusions in Treatment-Naïve Prostate Cancer Patients
Brief Title: Pharmacokinetics of IA and IV Ga68-PSMA-11 Infusion
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ryan Kohlbrenner, MD (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Sponsor-Investigator, Ryan Kohlbrenner, MD, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21921; NCI-2021-06580 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Prostate Adenocarcinoma; Prostate Carcinoma; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
Keywords: Ga68-PSMA-11
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Catheterization; gallium 68 PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ga-PSMA-11, PET/CT, Angiogram, and Prostatic Arterial Catheterization (Experimental): Patients receive 68Ga-PSMA-11 IV over 30 minutes and undergo dynamic PET imaging over infusion period and for 15 minutes after on day 1. One to 14 days later, patients undergo pelvic angiogram and prostatic arterial catheterization. Patients then receive 68Ga-PSMA-11 IA over 30 minutes and undergo dynamic PET imaging over infusion period and for 15 minutes after.
  Interventions: Procedure: Angiogram; Procedure: Catheterization; Drug: Gallium Ga-labeled PSMA-11; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Angiogram — Undergo angiogram
Procedure: Catheterization — Undergo prostatic arterial catheterization
Drug: Gallium Ga-labeled PSMA-11 — Given IV and IA
  Other Names: 68Ga-PSMA-11
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
Prostate-specific membrane antigen (PSMA) agents have shown promise in detecting and treating prostate cancer. Gallium-68-labeled PSMA-11 (68Ga-PSMA-11) is a radioactive agent that binds to prostate cancer cells and can be imaged using positron emission tomography (PET) scanners that detect radioactivity in the body. This early phase I study will use PET to determine if delivering 68Ga-PSMA-11 directly into the prostatic artery (intra-arterial (IA) administration) results in greater uptake in the prostate than delivering 68Ga-PSMA-11 into a vein in the arm (intravenous (IV) administration).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the maximum standardized uptake value (SUVmax) in tumoral regions-of-interest during prostatic arterial and intravenous 68Ga-PSMA-11 infusions.

SECONDARY OBJECTIVES:

I. To compare the tumoral time-activity curves for selective prostatic arterial and intravenous 68Ga-PSMA-11 infusions.

II. To study PSMA receptor saturation kinetics during selective prostatic arterial infusion of 68Ga-PSMA-11 (obtained only from arterial time activity curves [TACs] ipsilateral to the side of infusion).

OUTLINE:

Patients receive 68Ga-PSMA-11 IV over 30 minutes and undergo dynamic PET imaging over infusion period and for 15 minutes after on day 1. 1-14 days later, patients undergo pelvic angiogram and prostatic arterial catheterization. Patients then receive 68Ga-PSMA-11 IA over 30 minutes and undergo dynamic PET imaging over infusion period and for 15 minutes after.

After completion of study, patients are followed up with 24 hours after the IA infusion and PET scan.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years and less than or equal to 80 years.

  * Children are excluded from this study because the disease does not occur in children
  * Individuals from age 76 to age 80 must have a prior CT of the abdomen and pelvis within 5 years of first PSMA scan demonstrating non-occlusive pelvic atherosclerosis, regardless of smoking status
  * Individuals over the age of 80 are excluded from this study to improve the likelihood of a catheterizable prostatic artery, given the higher rates of occlusive atherosclerosis with advanced age
* Ability to provide informed consent
* Biopsy-proven unilateral or bilateral prostate adenocarcinoma, any stage (any N or any M)
* Large tumor burden, characterized by either

  * A discrete lesion with maximal tumor diameter >= 2.0cm on at least one affected side, documented on prostate magnetic resonance imaging (MRI) or Transrectal ultrasound (TRUS) within 4 months of first scan.
  * Infiltrative disease with primary pattern Gleason 4 adenocarcinoma in at least 4 of 6 sextant core biopsy locations on at least one affected side, documented in a surgical pathology report within 4 months of first scan.
* Gleason score >= 4+4
* Cancer of the Prostate Risk Assessment (CAPRA) score >= 6

Exclusion Criteria:

* Body mass index (BMI) > 35 kg/m^2
* Prior treatment for prostate cancer, or any use of anti-androgen therapy within 3 months of first scan
* History of any pelvic radiotherapy
* Severe atherosclerosis from prior CT imaging study, or greater than 10 pack-year smoking history if no prior imaging available.
* Stage IV or V chronic kidney disease by estimated glomerular filtration rate (eGFR) within 45 days of first scan
* Platelet count < 50 x 10^9/L and/or international normalized ratio > 1.5
* Severe allergy to iodinated contrast
* Active urinary tract infection or recent episode of prostatitis within 1 month of first scan
* Inability to tolerate prolonged supine positioning

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-03-22 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Maximum standardized uptake value (SUVmax) | Day 1 and from Day 2 up to Day 15 (2 days total)
  A two-sided paired t-test will determine whether the ipsilateral SUVmax values obtained during selective arterial 68Ga-PSMA-11 infusions are greater than those obtained during venous infusions. A similar paired analysis will be made during arterial infusions to compare tumoral regions of interest (ROIs) ipsilateral and contralateral to the side of the infusion. Means/medians, ranges/standard deviations will be calculated for each endpoint.

SECONDARY OUTCOMES:
Comparison of Mean SUV (SUVmean) | Day 1 and from Day 2 up to Day 15 (2 days total)
  Paired t-tests will determine whether SUVmean is different for intra-arterial (IA) time activity curves (TACs) when compared to intravenous (IV) TACs. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Time to SUVmax (TSUV) | Day 1 and from Day 2 up to Day 15 (2 days total)
  Paired t-tests will determine whether TSUV is different for IA TACs when compared to IV TACs. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Area under the curve (AUC) | Day 1 and from Day 2 up to Day 15 (2 days total)
  Paired t-tests will determine whether AUCs are different for IA TACs when compared to IV TACs. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Rate of 68Ga-PSMA-11 uptake | Day 1 and from Day 2 up to Day 15 (2 days total)
  To assess whether the rate of uptake is significantly different with selective arterial infusion, a two-sided paired t-test will compare the slopes for Selective arterial infusion, tumor ipsilateral to the side of radiotracer injection (IAIpsi) curves and Intravenous infusion, tumor ipsilateral to the side of corresponding arterial injection (IVIpsi) curves during each of the nine time intervals. Selective arterial infusion, tumor contralateral to the side of radiotracer injection (IACont) slopes will be similarly compared to those acquired from corresponding Intravenous infusion, tumor contralateral to the side of corresponding arterial injection (IVCont) data. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Time to early saturation effects | 1 day
  Specific to the IAIpsi TACs, the time to early saturation effects (Tese) will represent the time at which the second derivative of the curve becomes negative (i.e. when concavity in the curve is first noted). For the purposes of Tese, the aforementioned curve partitioning method will not be used. Descriptive statistics of Tese will be established, along with statistics for the corresponding mass dose administered (MDese) at Tese. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Mass dose at saturation | Day 1 and from Day 2 up to Day 15 (2 days total)
  Descriptive statistics of Tese will be established, along with statistics for the corresponding mass dose administered (MDese) at Tese. Means/medians, ranges/standard deviations will be calculated for each endpoint.
Comparison of Mean SUV during 15-minute washout (SUVwashout) | 1 day
  The mean SUVwashout and its standard deviation will be calculated for the 15-minute post-injection periods.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Kohlbrenner, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magnuska ZA, Roy R, Palmowski M, Kohlen M, Winkler BS, Pfeil T, Boor P, Schulz V, Krauss K, Stickeler E, Kiessling F. Combining Radiomics and Autoencoders to Distinguish Benign and Malignant Breast Tumors on US Images. Radiology. 2024 Sep;312(3):e232554. doi: 10.1148/radiol.232554. PMID 39254446
- [Derived] Kohlbrenner R, Wu X, Nguyen HG, Cooperberg MR, Chakravarty T, Carroll PR, Hope TA. Pharmacokinetic Comparison of Selective Prostatic Arterial and Intravenous PSMA PET/CT Radioligand Infusions in Primary Prostatic Adenocarcinoma. Radiology. 2024 Aug;312(2):e232544. doi: 10.1148/radiol.232544. PMID 39136560